CLINICAL TRIAL: NCT04435808
Title: Off Label Study to Evaluate the Efficacy of Hydroxychloroquine as Prophylaxis to Prevent Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection Among Health Care Workers at High Risk of Occupational Exposure to SARS-CoV-2
Brief Title: Efficacy of Hydroxychloroquine Prophylaxis for Health Care Workers at High Risk for COVID-19
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Stopped for futility by DSMB
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Walter Dehority, Associate Professor: Pediatrics Infectious Disease, University of New Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-206
Record Dates: First submitted 2020-06-04; First posted 2020-06-17 (Actual); Results first posted 2020-11-16 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine Arm (Experimental): Group A: up to 275 health care workers who choose to take hydroxychloroquine. Will receive a 600 mg loading dose, followed by 200 mg daily (tablets).
  Interventions: Drug: Hydroxychloroquine
- No Intervention Arm (No Intervention): Group B: Up to 75 health care workers who choose not to take hydroxychloroquine.

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine- oral administration: Duration: up to 90 days or until meeting study termination criteria. Subjects will recieve 600 mg loading dose, followed by 200 mg daily (tablets).
  Loading dose: 600 mg once for the first day Maintenance dose: 200 mg, daily
  Arms: Hydroxychloroquine Arm

SUMMARY:
The HCW Prophylaxis (HCWP) Study, single, open and off label intervention study. Up to 350 participants will be assigned to group that takes HCQ or group that opts to not take study medication. Participants will be UNM HEALTH SYSTEM HCW at high risk for occupational exposure to SARSCoV- 2. Study timepoints will include Day 1 screening/enrollment, 30 day, 60 day, and 90 day assessments. Questionnaires will be collected in all timepoints.

DETAILED DESCRIPTION:
This is an open and off label use, interventional, single site study. The HCWP Study eligibility are HCWs at high risk for SARS-CoV-2 exposure (eg MD/DO, NP, RN, and respiratory therapists in ED, Pediatric ED, Urgent Care, Pediatric Urgent Care and on Covid-19 units) at UNM HEALTH SYSTEM meeting all inclusion criteria. Total number of participants: 350 (Group A and B) Group A: up to 275 (HCW who choose to be provided HCQ). Will receive a 600 mg loading dose followed by 200 mg daily (tablets).

Group B: up to 75 (HCW who choose not to be provided HCQ)

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥18 years of age who are UNM HEALTH SYSTEM health care workers and are asymptomatic for known presenting symptoms of SARS-CoV-2:
2. UNMHS HCWs include: MD/DO, NP, RN, and respiratory therapists working in ED, Pediatric ED, Urgent Care, Pediatric Urgent Care or on Covid-19 units. Study PI's will consider study enrollment of HCWs from other settings, for example certain outpatient clinics or inpatient units.
3. Are not positive for SARS-CoV-2 testing
4. Willing and able to comply with survey completion, scheduled visits, treatment plan, and other study procedures
5. Willing and able to provide informed consent

Exclusion Criteria:

1. Known hypersensitivity to HCQ or other 4-aminoquinoline compounds
2. Currently hospitalized
3. Symptomatic with subjective fever, cough, or sore throat
4. Current medications exclude concomitant use of HCQ, for example anti-arrhythmic agents, digoxin, cyclosporin, cimetidine, or tamoxifen.
5. Concomitant use of other anti-malarial treatment or chemoprophylaxis
6. History of retinopathy of any etiology
7. Psoriasis
8. Porphyria
9. Known bone marrow disorders with significant neutropenia (polymorphonuclear leukocytes <1500) or thrombocytopenia (<100K)
10. Known liver disease
11. Known long QT syndrome
12. Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of the study drugs or planned use during the study period. There may be some exceptions to requiring a 30-day washout that will be evaluated by the Co-Investigators on a case by case basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxychloroquine Arm: Group A: 0 health care workers who chose to take hydroxychloroquine
  Hydroxychloroquine: Hydroxychloroquine- oral administration: Duration: up to 90 days or until meeting study termination criteria.
  Loading dose: 600 mg once for the first day Maintenance dose: 200 mg, daily
- No Intervention Arm: Group B: 1 health care worker who chose not to take hydroxychloroquine
Period: Overall Study
Arm/Group | Hydroxychloroquine Arm | No Intervention Arm
Started | 0 | 1
Completed | 0 | 0 (Study stopped prior to any data collection for this lone participant)
Not Completed | 0 | 1
Not completed — Study stopped by DSMB | 0 | 1

BASELINE CHARACTERISTICS:
Population: DSMB stopped the study
Groups:
- Hydroxychloroquine Arm: Group A: 0 health care workers who choose to take hydroxychloroquine
  Hydroxychloroquine: Hydroxychloroquine- oral administration: Duration: up to 90 days or until meeting study termination criteria.
  Loading dose: 600 mg once for the first day Maintenance dose: 200 mg, daily
- No Intervention Arm: Group B: 1 health care workers who chose not to take hydroxychloroquine
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine Arm | No Intervention Arm | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: SARS-CoV-2 Infection
Description: Number of health care workers who become infected with SARS-CoV-2 as detected by PCR
Time Frame: 3 months
Population: DSMB stopped trial early prior to any data collection.
Arm/Group | Hydroxychloroquine Arm | No Intervention Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Not collected
Description: Not collected
Groups:
- No Intervention Arm: Group B: 0 health care worker who chose not to take hydroxychloroquine
Arm/Group | Hydroxychloroquine Arm | No Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT04435808/Prot_SAP_001.pdf
  • Informed Consent Form (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT04435808/ICF_000.pdf